CLINICAL TRIAL: NCT02827409
Title: A Randomized Controlled Trial of Short-Delay Cord Clamping as Compared to Extended- Delayed Cord Clamping in Term Neonates That Require Resuscitation.
Brief Title: Short-Delay Cord Clamping Compared to Extended- Delay Cord Clamping in Term Neonates That Require Resuscitation.
Acronym: Term-NRIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anup Katheria, M.D. (Other)
Responsible Party: Sponsor-Investigator, Anup Katheria, M.D., Director Neonatal Reseach Institute, Sharp HealthCare
Organization: Sharp HealthCare (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Term-NRIC
Record Dates: First submitted 2016-07-05; First posted 2016-07-11 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Placental Transfusion
Keywords: Delayed cord clamping
MeSH Terms: conditions — Fetofetal Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short Delay Cord Clamping (Active Comparator): Subject will have umbilical cord clamped and cut by 1 minute of life.
  Interventions: Procedure: Short Delay Cord Clamping
- Extended Delay Cord Clamping (Active Comparator): Subject will have umbilical cord clamped and cut after at least 5 minutes of delayed cord clamping. Duration of cord clamping after 5 minutes will depend on if the subject is breathing and/or if the cord has stopped pulsating
  Interventions: Procedure: Extended Delay Cord Clamping

INTERVENTIONS:
Procedure: Short Delay Cord Clamping — Delay cord clamping will occur for up to 1 minute. Subject will be placed on mother's abdomen for warmth and stimulation. If the subject is depressed they will be transferred to the radiant warmer for resuscitation.
  Arms: Short Delay Cord Clamping
Procedure: Extended Delay Cord Clamping — Extended delay cord clamping will occur for at least 5 minutes and will continue until the subjects begins breathing and/or the cord stops pulsating. Subject will be placed on mother's abdomen for warmth and stimulation. If the subject is depressed they will be transferred to the LifeStart bed for resuscitation adjacent to the mother's bedside.
  Arms: Extended Delay Cord Clamping

SUMMARY:
To determine whether performing extended delayed cord clamping in term neonates that require resuscitation improves early transition as compared to short-delayed cord clamping.

DETAILED DESCRIPTION:
All subjects will receive delayed cord clamping. One group (short-delay) will receive up to one minute of delayed cord clamping and then will be placed either on the mother's abdomen or the life-start trolley if extensive resuscitation is required.

The second group will receive delayed cord clamping for at least 5 minutes and continue until the baby has established breathing without additional support or is stable on respiratory support (no longer received mask PPV for at least 1-2 minutes, i.e. stable on CPAP or intubated). The subject will initially be placed on the mother's abdomen or if the subject needs extensive resuscitation they will be moved to the LifeStart bed to receive resuscitation measures.

In either group if the baby is deemed to be unstable (by medical team) to be on the life-start trolley the cord will be clamped and the baby will be moved to an adjacent warmer for resuscitation.

ELIGIBILITY:
* Inclusion Criteria: Gestation 37 weeks or greater that require attendance at delivery of neonatal provider due to an at risk delivery.
* Exclusion Criteria: Planned cesarean birth, placental abruption, multiple gestations, or known congenital anomalies.

Ages: 37 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2016-07; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Cerebral tissue oxygenation | 12 hours of life
  The need for oxygen, positive pressure ventilation, intubation

SECONDARY OUTCOMES:
Heart rate | First 5 minutes of life
  Heart rate obtained by pulse doppler, EKG, oximetry or a combination of all
Oxygen saturation | over the first 5 minutes of life
  data will be averaged over each minute of life
delivery room resuscitation | at birth
  did the infant require resuscitation such as stimulation to breathe, oxygen, positive pressure ventilation etc.
Blood pressure | 12 hours of life
Hemoglobin | First 5 minutes of life
  if Hemoglobin oximeter available
Hemoglobin | 12 hours of life
  if Hemoglobin oximeter available
Apgar Score | First 10 minutes of life
  1, 5 and 10 minute Apgar
Arterial and Venous Umbilical Cord Blood Gases | At birth
Need for NICU admission | at birth
Need for hypothermia for hypoxic ischemic encepalopathy | at birth
  will be assessed by primary physician using defined criteria for hypothermia
Hospitalization days | up to 24 weeks
Bilirubin level | 12-48 hours
  by transcutaneous or serum if available. percentile on curve will be document to adjust for different time frames.
Neurodevelopmental impairment | 12 month followup
  by Ages and Stages questionnaire or Bayley 3scales of infant and toddler development
Post delivery survey | at birth
  Survey of practitioners (LD nurse, OB, neonatal team) about procedure

CONTACTS AND LOCATIONS:
Overall Officials: Anup Katheria, MD, Principal Investigator — Sharp HealthCare
Locations (1):
- Sharp Mary Birch Hospital for Women and Newborns, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
small pilot study of term infants

REFERENCES:
- [Derived] Katheria AC, Brown MK, Faksh A, Hassen KO, Rich W, Lazarus D, Steen J, Daneshmand SS, Finer NN. Delayed Cord Clamping in Newborns Born at Term at Risk for Resuscitation: A Feasibility Randomized Clinical Trial. J Pediatr. 2017 Aug;187:313-317.e1. doi: 10.1016/j.jpeds.2017.04.033. Epub 2017 May 16. PMID 28526223